CLINICAL TRIAL: NCT00136188
Title: Role of NO Activity for the Development of Diabetic Nephropathy
Brief Title: Nitric Oxide (NO) Activity and Diabetic Nephropathy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: SFB 423 TP B5
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Diabetic Nephropathies
Keywords: Prediabetes; Metabolic Syndrome; Healthy Controls; Endothelial function
MeSH Terms: conditions — Diabetic Nephropathies; Prediabetic State; Metabolic Syndrome | interventions — Folic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Folic Acid — oral administration of folic acid 5mg /d for 4 weeks

SUMMARY:
Experimental data suggest that oxidative stress and endothelial dysfunction are key players in the pathogenesis of diabetic nephropathy. In the last few years the investigators were able to establish a method to assess endothelial function of the renal vasculature in humans and started to systematically study a variety of cardiovascular disorders known to be associated with endothelial dysfunction in other vascular beds, including hypertension, hypercholesterolemia and type-2 diabetes. In patients with type-2 diabetes the investigators could demonstrate that despite unaltered basal and stimulated NO-activity, the renal response to the antioxidant vitamin C was more pronounced compared to control subjects. These data suggest that oxidative stress is increased in the renal vasculature of diabetic patients. Furthermore, NO-activity in diabetic patients appears to be upregulated to compensate for the increase in oxidative stress. This hypothesis is supported by the demonstration of increased endothelial nitric oxide synthase (eNOS) expression in kidney biopsies of diabetic patients.

The major focus of the investigators' current research activities is to assess the role of endothelial dysfunction in the very early stages of diabetic nephropathy. To this end, patients with increased fasting glucose or metabolic syndrome will be studied in comparison with an age-matched control group. Endothelial function and the role of oxidative stress will be assessed in the renal vasculature in all groups. In parallel, the investigators will study endothelial function in the forearm by venous occlusion plethysmography and in the retinal vasculature by scanning laser doppler flowmetry to dissect regional differences in the regulation of endothelial function. Further aspects include the role of microalbuminuria, glomerular hyperfiltration, and endogenous inhibitors of NO synthase such as NG,NG-Dimethyl-L-Arginine (ADMA). In a therapeutic approach, the investigators will determine the effects of various antioxidant treatment strategies on endothelial function and their potential role in the prevention of diabetic nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18-65 with diabetes, prediabetes or metabolic syndrome
* Male and female healthy control subjects aged 18-65

Exclusion Criteria:

* Advanced damage of vital organs (grade III and IV retinopathy)
* Therapy with a not approved concomitant medication in the last 4 weeks prior to intake of the first trial medication, especially lipid lowering and antidiabetic medications (washout phase)
* Blood donation within the last 4 weeks
* Patients with arterial fibrillation or atrioventricular (AV)-block (II and more)
* Patients with anamnestic myocardial infarct
* Patients with depression
* Patients with seizure disorders
* Patients with unstable angina pectoris including electrocardiogram (ECG)-aberrations or cardiac insufficiency New York Heart Association (NYHA) Stadium III and IV
* History of a malignant illness with the exception of those patients who have recovered for more than 10 years or have a basalioma of the skin.
* Actual or anamnestic alcohol or drug abuse
* History of organ transplant
* Anaphylaxis or known therapy resistance to any of the used test matters.
* Therapy with a not approved concomitant therapy
* Participation in another study within three months prior to study inclusion
* Illnesses, which can influence the pharmacodynamics or pharmacokinetics of the test substance
* Liver or kidney diseases; SGOT, GPT, γ-GT, AP, bilirubin and creatinine above 200% of standard
* Patients who are not sufficiently compliant, or patients who are not capable or willing to appear for controlling visits
* Severe or unstable medical or psychiatric illnesses, which will, in the estimation of the examiner, endanger the safety of the proband or the successful participation in the study
* Presumed risk of transmission of HIV or hepatitis via blood from the proband

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change in renal endothelial function | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Roland E Schmieder, MD, Principal Investigator — CRC, Medizinische Klnik 4 - Nephrology and Hypertension, Uni Erlangen-Nürnberg; Markus P Schlaich, MD, Principal Investigator — CRC, Medizinische Klnik 4 - Nephrology and Hypertension, Uni Erlangen-Nürnberg
Locations (1):
- CRC, Medizinische Klnik 4 - Nephrology and Hypertension, Uni Erlangen-Nürnberg, Erlangen, Germany

REFERENCES:
- [Derived] Kannenkeril D, Bosch A, Harazny J, Karg M, Jung S, Ott C, Schmieder RE. Early vascular parameters in the micro- and macrocirculation in type 2 diabetes. Cardiovasc Diabetol. 2018 Sep 19;17(1):128. doi: 10.1186/s12933-018-0770-4. PMID 30231923
- [Derived] Ott C, Schneider MP, Delles C, Schlaich MP, Schmieder RE. Reduction in basal nitric oxide activity causes albuminuria. Diabetes. 2011 Feb;60(2):572-6. doi: 10.2337/db09-1630. PMID 21270268